CLINICAL TRIAL: NCT05427396
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability,of Recombinant Humanized Anti-BTLA Monoclonal Antibody (JS004) Injection Combined Witht Oripalimab in Patients With Advanced Solid Tumors
Brief Title: A Phase I Clinical Study of Recombinant Humanized Anti-BTLA Monoclonal Antibody (JS004) Injection Combined With Toripalimab Injection in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was stopped early on the initiative of the sponsor on the basis of a change in the research and development strategy without safety concerns
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS004-005-I
Record Dates: First submitted 2022-06-05; First posted 2022-06-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Liver Cancer, Esophageal Squamous Cell Carcinoma, Gastric Adenocarcinoma, Cervical Cancer, MSI-H Colorectal Cancer
MeSH Terms: conditions — Liver Neoplasms; Esophageal Squamous Cell Carcinoma; Uterine Cervical Neoplasms | interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS004 200 mg in combination with Toripalimab Injection 240 mg was administered every 3 weeks (Other)
  Interventions: Drug: JS004; Drug: Toripalimab Injection

INTERVENTIONS:
Drug: JS004 — Usage and dosage: Inject 200mg once every 3 weeks
Drug: Toripalimab Injection — Usage and dosage: Inject 240mg once every 3 weeks

SUMMARY:
This is an open-label phase I study to evaluate the safety, tolerability, and initial efficacy of JS004 injection combined with Toripalimab Injection in patients with advanced solid tumors who have failed standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily;
2. Patient (both sex) ≥ 18 and ≤70 years at the time of signing informed consent;
3. Expected survival ≥ 3 months;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
5. Patients with advanced solid tumors confirmed histologically or cytologically
6. At least one measurable lesion as a target lesion (RECIST v1.1 criteria);
7. Agree to provide tumor tissue samples (provide fresh biopsy samples before treatment as far as possible;
8. The patient has good organ function as indicated by screening laboratory results
9. Males of reproductive potential or females of childbearing potential must use effective contraceptive methods (such as oral contraceptives, intrauterine device or barrier method combined with spermicide) during the trial and continue contraception for 6 months after the end of treatment;
10. Good compliance and cooperated with the follow-up.

Exclusion Criteria:

1. Any malignancy other than the disease under study within the past 5 years, except for malignancies that can be expected to be cured after treatment (including but not limited to adequately treated thyroid cancer, carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated surgically with curative intent);
2. patients received systemic antitumor therapy (including chemotherapy, small-molecule targeted drug therapy, endocrine therapy, etc.) or local antitumor therapy within 4 weeks prior to 1st administration
3. Received immunotherapy (including antibody and cell therapy) within 4 weeks prior to 1st administration
4. Received allogeneic hematopoietic stem cell transplantation or solid organ transplantation in the past;
5. Central nervous system metastases and/or cancerous meningitis
6. Have or are suspected of having active autoimmune diseases, including but not limited to systemic lupus erythematosus rheumatoid arthritis inflammatory bowel disease autoimmune hepatitis
7. A large amount of hydrothorax or ascites or pericardial effusion with clinical symptoms or requiring symptomatic treatment;
8. Have serious cardiovascular and cerebrovascular diseases, such as poorly controlled hypertension (systolic blood pressure>140mmHg and/or diastolic pressure> 90mmHg) or pulmonary arterial hypertension; Unstable angina or had a myocardial infarction in the 6 months prior to study use and had coronary artery bypass grafting or stenting; Chronic heart failure with grade 2 heart function (NYHA); Degree above heart block; Left ventricular ejection fraction (LVEF)<50%; Cerebrovascular accident (CVA) or transient ischemic attack (TIA) occurred within 6 months prior to medication
9. Pulmonary disease: interstitial pneumonia, obstructive pulmonary disease and symptomatic bronchospasm;
10. A positive result for human immunodeficiency virus (HIV) antibody test;
11. Known active tuberculosis (TB).
12. Live vaccine was administered within 4 weeks prior to 1st administration
13. Major surgical procedures (as defined by the investigator, e.g., open biopsy, severe trauma, etc.) within 4 weeks prior to 1st administration
14. Have a history of psychotropic drug abuse and unable to withdraw or have mental disorders;
15. Pregnant or lactating woman;
16. Known to be allergic to JS004 or toripalimab and its components;
17. Other severe, acute or chronic medical or psychiatric disorders or laboratory abnormalities that, in the investigator's opinion, may increase the risk associated with study participation or may interfere with the interpretation of study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events (AE) and serious adverse events (SAE) were assessed | 2 years
  Incidence and severity of adverse events (AE) and serious adverse events (SAE) as assessed according to NCI-CTCAE 5.0, as well as abnormalities in vital signs, electrocardiogram, and laboratory tests

SECONDARY OUTCOMES:
OS | 2 years
  Duration of Response
DOR | 2 years
  Duration of Response
DCR | 2 years
  Disease Control Rate
PFS | 2 years
  Progression-free survival
ORR | 2 years
  Overall Response Rate
TTR | 2 years
  Time to remission
TTP | 2 years
  time to progression

OTHER OUTCOMES:
ORR | 2 years
  Objective response rate based on iRECIST criteria (Version 2017);
DOR | 2 years
  duration of response based on iRECIST criteria (Version 2017);
DCR | 2 years
  disease control rate based on iRECIST criteria (Version 2017);
PFS | 2 years
  progression-free survival based on iRECIST criteria (Version 2017);

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No